## Minimum Informed Volunteer Consent Form (Sample)

This study was carried out by Ebrar ATAK (PT. Msc.) prepared the doctorate program of Istanbul Medipol University Institute of Health Sciences Physiotherapy and Rehabilitation as a thesis study and approved by Istanbul Medipol University Non-Clinical Studies Ethics Committee. The aim of this study is to determine the effect of dual-task balance training on cognitive functions and to evaluate its effectiveness. Participation in the study should be on a voluntary basis. In the study, no personally identifiable information is required from you. The data obtained in the study will be kept strictly confidential and evaluated only by the researchers; The information obtained will be used in scientific publications.

Persons who can participate in the planned physiotherapy program will be included in the study. However, if you feel uncomfortable with the program or any other reason during the participation, you are free to interrupt and quit. In such a case, it is sufficient to tell the person who applies the physiotherapy program that you cannot complete the program. At the end of the study, your questions will be answered. Thank you in advance for participating in this study. For more information about the study, see Exp. PT. You can get detailed information by contacting Ebrar ATAK (05052049391).

I participate fully in this effort voluntarily and I know that I can interrupt at any time. I agree to the use of the information and data obtained in scientific publications. (Fill out and sign the form and return it to the practitioner).

| Name Surname | Date | 2 | Signature |
|--------------|------|-----|-----------|
| _ | / | - / | |